CLINICAL TRIAL: NCT07160101
Title: "Comparative Efficacy Of Eggshell Derived Nano Hydroxyapatite Over Hydroxyapatite In The Treatment Of Periodontal Intrabony Defects: A Clinico-Radiographic Study"
Brief Title: Comparison of Effects of Eggshell Derived Nano Hydroxyapatite and Hydroxyapatite in Management of Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr R Viswa Chandra (Other)
Responsible Party: Sponsor-Investigator, Dr R Viswa Chandra, PROFFESSOR AND HEAD OF THE DEPARTMENT, SVS Institute of Dental Sciences
Organization: SVS Institute of Dental Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/1/2022
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Periodontal Intrabony Defects; Bone Regeneration
MeSH Terms: interventions — Durapatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group Eggshell derived nano hydroxyapatite (Experimental): In Test group after flap reflection & degranulation, bone graft i.e Eggshell derived nano hydroxyapatite is placed into defect.
  Interventions: Other: Eggshell derived nano hydroxyapatite
- Control group (Active Comparator): In Control group, after flap reflection & debridment bone graft i.e Hydroxyapatite is placed into defect.
  Interventions: Other: Hydroxyapatite

INTERVENTIONS:
Other: Eggshell derived nano hydroxyapatite — Eggshell derived nano hydroxyapatite has high solubility and allows faster integration & replaces with osseous tissue
  Arms: Test group Eggshell derived nano hydroxyapatite
Other: Hydroxyapatite — Hydroxyapatite has similar chemical composition with crystalline structure of native bone
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate osseous regenerative efficacy of eggshell derived nanohydroxyapatite in comparison with hydroxyapatite The test group includes patients with intrabony defects where flap surgery will be performed & Eggshell derived nano hydroxyapatite (ESnHA) is placed.

DETAILED DESCRIPTION:
Experimental : Main treatment group Eggshell derived nano hydroxyapatite is placed into defect site Comparator : In patients allocated to control group, only Hydroxyapatite is placed.

ELIGIBILITY:
Inclusion Criteria:

Presence of Two-walled or three-walled intrabony defects & Probing pocket depths (PPD) of >5mm after initial therapy Systemically healthy male and female patients of age >18 years

Exclusion Criteria:

Medically compromised patients Pregnant women, Heavy smokers, and Patients who underwent radiotherapy or chemotherapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
RVG | 3months & 6months
  Radiovisiography will be used to assess bone regeneration achieved post operatively
Probing Depth | 3 months & 6months
Clinical Attachment Level | 3 months & 6 months

SECONDARY OUTCOMES:
Full mouth Plaque index | 3 months & 6 months
  Full mouth plaque index was measured using Turesky modification of the Quigley-Hein Index at baseline, 3 months and 6 months
Full mouth Gingival index | 3 months & 6 months
  Full mouth gingival index was measured using Loe & Silness Index at baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Svs Institute of Dental Sciences, Mahbūbnagar, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided